CLINICAL TRIAL: NCT07260578
Title: Safety and Efficacy of Ellacor Micro-coring Following Best Practices on Technique and Post-Procedural Care
Brief Title: Safety and Efficacy of Ellacor® Micro-coring® Following Best Practices on Technique and Post-Procedural Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TP-00456
Record Dates: First submitted 2025-11-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Best Practices; Ellacor; Micro-coring Post Care; Ellacor Post Care
Keywords: ellacor post care; micro-coring best practices; ellacor best practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Regenerating Skin Nectar (by Alastin) + Tegaderm (Active Comparator): Alastin to be applied post procedure followed up Tegaderm. Tegaderm will be left on for 12 hours. Alastin will be applied twice daily for the duration of the study
  Interventions: Device: ellacor Micro-Coring Technology
- Kerra+ Recovery Cream (by Quthero) + Tegaderm (Active Comparator): Patients will receive Kerra+ post procedure followed by Tegaderm. The Tegaderm is removed after 12 hours. Kerra+ will be applied twice daily for the duration of the study.
  Interventions: Device: ellacor Micro-Coring Technology
- Ariessence Platelet-Derived Growth Factor (PDGF) solution +Alastin + Tegaderm (Active Comparator): Patients will receive PDGF immediately post procedure followed by Alastin followed by Tegaderm. The Tegaderm will be removed after 12 hours and the Alastin will continue to be applied twice daily for the duration of the study
  Interventions: Device: ellacor Micro-Coring Technology
- Ariessence PDGF solution + Kerra+ Recovery Cream + Tegaderm (Active Comparator): Patients will receive PDGF immediately post procedure followed by Kerra+ followed by Tegaderm. The Tegaderm will be removed after 12 hours and the Kerra+ will continue to be applied twice daily for the duration of the study
  Interventions: Device: ellacor Micro-Coring Technology
- Tegaderm Only (Active Comparator): Patient will only receive Tegaderm for post-care
  Interventions: Device: ellacor Micro-Coring Technology

INTERVENTIONS:
Device: ellacor Micro-Coring Technology — ellacor will be used to treat moderate-severe wrinkles in the mid to lower face in subjects aged between 45-65.
  Other Names: ellacor; micro-coring; dermal micro-coring

SUMMARY:
Since its inception of being marketed in the United States in 2021, physicians have used various post procedure skin care regimen to facilitate recovery. This study aims to examine the use of three post care products in five skin care regimens

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult, between the ages of 45 and 65
2. Fitzpatrick Skin Type I to IV
3. Have moderate to severe wrinkles on the mid and lower face, according to Lemperle Wrinkle Severity Scale (LWSS), i.e. score 3, 4 or 5.
4. Willingness to sign Informed Consent Form

Exclusion Criteria:

1. Pregnant women or nursing mothers
2. Patients with dermatosis, open wounds, sores, or irritated skin in the treatment area
3. Patients with allergy to stainless steel or to topical, oral, or injected medications or preparations that may be used during the procedure, such as petrolatum, lidocaine, bupivacaine, chlorhexidine, or povidone-iodine
4. Patients with a history or presence of any clinically significant bleeding disorder

i. Patients with dermatological or autoimmune conditions that may affect the treatment outcome; these may include, but are not limited to: actinic keratosis, raised nevi, rosacea, melasma, active acne, cutaneous papules/nodules, active inflammatory lesions, dermatitis, psoriasis, cellulitis, urticarial folliculitis, acute inflammatory phase of scleroderma, rheumatoid arthritis, eczema, psoriasis, allergic dermatitis, collagen disorders, or lupus e. Patients with systemic infections or acute local skin infections (as Hepatitis disorders type A, B, C, D, E or F or HIV infection) f. Patients who are on a high dose of anti-coagulants or blood-thinning substances, e.g., aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), warfarin, heparin, acetylsalicylic acid during the previous fourteen (14) days g. Patients who are on courses of chemotherapy, high-dose corticosteroid use, or radiation in the treatment area h. Patients have undergone plastic surgery of the face within the last twelve (12) months or have any facial surgical scars less than twelve (12) months old i. Patients who have undergone injections of dermal fillers, fat, or botulinum toxin, as well as any minimally invasive/invasive skin treatment in the treatment area during the previous six (6) months j. Patients with scars less than six (6) months old in the treatment area k. During the study time frame, unwilling to refrain from receiving these following aesthetic treatments: toxin, filler, any skin resurfacing (laser, RF, ultrasound, microneedling, etc.); l. Have enrolled in another clinical trial during or overlapping part of this study m. Unwilling to have facial photography taken for the study purpose n. Any physical or psychological factors, in the judgment of the study investigator, may prevent subject from performing the procedure correctly.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) | GAIS Assessment will be performed under a timeframe of 90 days
  Treatment improvement will be evaluated based off the 7 grade GAIS by both the subject and the physician.

SECONDARY OUTCOMES:
Clinical Assessment | Clinical assessment will be performed at each follow up throughout the study period.
  Clinical assessment will be performed, and graded on a 0-3 scale on Day 0, Day 7, Day 30, and Day 90- 0 = absent, 1 = mild, 2 = moderate, 3 = severe for the following side effects:
  * Bleeding
  * Erythema - redness
  * Ecchymosis - bruising
  * Dryness, roughness
  * Crusting Tenderness
  * Numbness
  * Edema - swelling
  * Burning
  * Tightness/Pulling of Skin
  * Pain/Discomfort
  * Tingling
  * Skin Peeling
  * Circular Marks on skin
  * Any other observation

OTHER OUTCOMES:
Safety Outcomes | Day 0 to end of study period
  Safety will be evaluated throughout the duration of the study by recording adverse events on Day 0, Day 7, Day 30, and Day 90
Subject Satisfaction Survey | Day 90
  Subject satisfaction data will be collected via a written questionnaire at the 90-day post procedure final follow-up visit. This questionnaire will be composed of 5-point Likert scale questions, as well as free-text responses. Subjects will be asked to determine overall satisfaction with the treatment. The choices will be: 1) very unsatisfied; 2) somewhat unsatisfied; 3) neither unsatisfied nor satisfied; 4) somewhat satisfied; 5) very satisfied.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami Dermatology And Laser Institute, Miami, Florida
  - Caloaesthetics Plastic Surgery Center, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No